CLINICAL TRIAL: NCT05618756
Title: Effects of Acute Cannabidiol (CBD) Supplementation on Nutrient Metabolism and Energy Intake in Healthy Adults
Brief Title: CBD, Nutrient Metabolism and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Lewis James, Senior Lecturer in Nutrition, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 5553
Record Dates: First submitted 2022-02-23; First posted 2022-11-16 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus); Lipid Metabolism Disorders; Appetitive Behavior
MeSH Terms: conditions — Glucose Metabolism Disorders; Lipid Metabolism Disorders; Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (Experimental): 300 mg CBD (KannaSwiss, Kölliken, Switzerland) dissolved in 1 ml hemp oil. Provided orally in gelatin capsules.
  Interventions: Dietary Supplement: Acute oral CBD supplementation
- Placebo (Placebo Comparator): 1 ml hemp oil. Provided orally in gelatin capsules.
  Interventions: Dietary Supplement: Acute oral placebo supplementation

INTERVENTIONS:
Dietary Supplement: Acute oral CBD supplementation — 1 ml hemp oil containing 300 mg CBD, within gelatin capsules, ingested orally.
  Arms: Cannabidiol
Dietary Supplement: Acute oral placebo supplementation — 1 ml hemp oil containing no CBD, within gelatin capsules, ingested orally.
  Arms: Placebo

SUMMARY:
CBD may affect metabolic control and energy intake. However, there is currently little data regarding these specific outcomes in humans. Therefore, this study will investigate whether a single 300 mg dose of CBD can improve metabolic control following a meal and/or reduce energy intake at a subsequent meal. Healthy, adult volunteers will complete two conditions in a crossover design, comparing outcomes following both CBD and placebo supplementation.

ELIGIBILITY:
Inclusion Criteria:

• Self-report as healthy, male or female, aged 18-50, body mass index ≥18.5 and <30.0

Exclusion Criteria:

* Currently engage in >10 hours moderate or vigorous intensity physical activity per week
* Have consumed CBD or cannabis at all within the past two months
* Have used CBD or cannabis regularly (>2x in a week) within the past four months
* Are suffering from any clinically significant illness
* Have regularly used tobacco within the previous 6 months (> 2/week)
* Currently use any prescription or over-the-counter medications (except for hormonal contraception and simple painkillers)
* Have given a standard blood donation within 30 days of screening
* Are currently pregnant or lactating
* Are allergic/intolerant to any ingredients in food items provided during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Energy intake | ~5-30 minutes (time taken to eat a single meal)
  Self-selected energy intake at an ad libitum mixed meal
Postprandial Glycaemia | 3 hours
  Plasma glucose response to a mixed meal (plasma glucose concentrations and area under curve)
Postprandial Triglyceridaemia | 3 hours
  Plasma triglyceride response to a mixed meal (plasma triglyceride concentrations and area under curve)

SECONDARY OUTCOMES:
Postprandial Insulinaemia | 3 hours
  Plasma Insulin response to a mixed meal (plasma insulin concentrations and area under curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No